CLINICAL TRIAL: NCT02668809
Title: Iowa Nursing Facility Oral Hygiene Intervention: A Pilot Study
Brief Title: Oral Hygiene Intervention Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leonardo Marchini (Other)
Collaborators: Ivoclar Vivadent AG (Industry); Delta Dental of Iowa (Other)
Responsible Party: Sponsor-Investigator, Leonardo Marchini, DDS, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: INFOH
Record Dates: First submitted 2016-01-22; First posted 2016-01-29 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Dental Caries; Gingivitis
MeSH Terms: conditions — Dental Caries; Gingivitis | interventions — Surveys and Questionnaires; Consent Forms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Experimental Group 1 (Experimental): consent, oral health assessment, questionnaires, Educational Program, clinical exam, microbiological sampling, monitoring adherence.
  Interventions: Other: oral health assessment; Other: Questionnaires; Other: Clinical Exam; Other: Microbiological sampling; Other: Monitoring Adherence; Other: Consent; Other: Educational Program
- Experimental group 2 (Experimental): Consent, oral health assessment, questionnaires, Educational Program, clinical exam, microbiological sampling, monitoring adherence, varnish application
  Interventions: Other: oral health assessment; Other: Questionnaires; Other: Clinical Exam; Other: Microbiological sampling; Other: Monitoring Adherence; Other: Varnish application; Other: Consent; Other: Educational Program
- Control Group (Placebo Comparator): Consent,clinical exam, microbiological sampling, questionnaires
  Interventions: Other: oral health assessment; Other: Questionnaires; Other: Clinical Exam; Other: Microbiological sampling; Other: Consent

INTERVENTIONS:
Other: oral health assessment — A baseline oral health assessment of both residents and direct care workers will be conducted before interventions are initiated. Data will be entered directly into a spreadsheet format using the chairside software program to be developed as part of this proposal.
Other: Questionnaires — Age, sex, race, nutrition (mini-nutri), quality of life (SF-36), OHIP-14, GOHAI, sources of payment for the NF residency, comorbid conditions (e.g., constipation, arthritis), weight, medications, cognitive status (mini-mental) , dry mouth sensation, x-ray documented pneumonia;
Other: Clinical Exam — Dentate status, dental/denture plaque index, DMFS (including root surfaces), gingival bleeding index, plaque index, presence of oral lesions, verification of mouth dryness;
Other: Microbiological sampling — Samples will be collected by swabbing patients intra-oral tissues. Samples will be separately collected from dentures and oral tissues for edentulous patients, also using swabs. All samples will be suspended in saline solution.
Other: Monitoring Adherence — Adherence to the protocol will be evaluated through unannounced observations at the NF by study personnel twice per month. Adherence is determined by direct observation of the DCW administering the intervention.
  Arms: Experimental Group 1; Experimental group 2
Other: Varnish application — 1% chlorhexidine varnish application group" will receive the educational program described above. In addition, residents who need supervision or are unable to perform oral hygiene procedures will receive 1% chlorhexidine varnish application monthly by the dental hygienist. No additional time commitment will be necessary.The direct care workers will NOT receive any varnish.
  Arms: Experimental group 2
Other: Consent — Both the residents and primary care workers will be asked to participate on the study, and the investigators will provide information and collect signed informed consents primarily during two in person visits to each nursing facilities.
Other: Educational Program — Cognitively capable residents will receive instruction on how to perform their own oral hygiene accordingly to their own needs; and 2) Direct care workers will receive instruction on how to perform oral hygiene for dependent residents or supervise the oral hygiene routines of independent patients. For both 1) and 2) above, dental hygienists will provide a short, standardized presentation and hands-on demonstration.
  Arms: Experimental Group 1; Experimental group 2

SUMMARY:
The main goals of this pilot study are to develop a nursing home-customized oral hygiene protocol, intended to be delivered primarily by dental hygienists and primary care providers, and to identify potential obstacles and barriers to overcome in designing a subsequent definitive study on the same topic.

DETAILED DESCRIPTION:
For the purposes of this pilot study, a convenience sample from six (6) to twelve (12) nursing facilities will be selected and randomly assigned into three groups: Experimental group 1 (educational program only, performed by a dental hygienist); Experimental group 2 (educational program plus 1% chlorhexidine varnish application monthly for the residents); Control group (current oral hygiene practice). Several objective and subjective oral and general health measures will be observed before and after the interventions to evaluate the impact of the interventions on the oral and general health of the residents and also of the direct care workers.

Assigned personnel in each nursing facility (NF) will be interviewed to identify possible barriers to provide oral care. Each interview will take one hour, approximately.

All residents that agree to participate will be interviewed and have an oral examination and dental plaque sample collection by the investigators. Each appointment will take 30 minutes. The subject's health record in the nursing facilities will be abstracted for medical information (date of birth, sex, race, source of payment for NF residency, comorbid conditions, weight, height, medications, number of febrile days, and x-ray documented pneumonia episodes).

After that, the educational program will be delivered in a standardized fashion for all NF in the "educational program only group": 1) Cognitively capable residents will receive instruction on how to perform their own oral hygiene accordingly to their own needs (approximately 15 minutes); and 2) Direct care workers will receive instruction on how to perform oral hygiene for dependent residents or supervise the oral hygiene routines of independent patients (01 hour session). For both 1) and 2) above, dental hygienists will provide a short, standardized presentation and hands-on demonstration. In addition, the dental hygienist will provide in situ oral care (plaque and gingival bleeding index assessment, microbiological sampling and toothbrushing with chlorhexidine mouth rinse) on a bi-weekly basis during the study period (15 minute each appointment) .

The "educational program plus 1% chlorhexidine varnish application group" will receive the educational program described above. In addition, residents who need supervision or are unable to perform oral hygiene procedures will receive 1% chlorhexidine varnish application monthly by the dental hygienist. No additional time commitment will be necessary.The direct care workers will NOT receive any varnish.

The control group will not receive any intervention through this protocol during the formal study period, but if the initial results are promising they will be invited after the formal study period to receive the educational program.

After a six month period from the initial examination,all residents and direct care workers that agree to participate will be interviewed and have an oral examination and dental plaque sample collection by the investigators again. Each appointment will take 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* be a resident or primary care worker in one of the following nursing homes: Linn Manor Care Center Simpson Memorial Home, Inc., Wilton Retirement Community, All-American Care of Muscatine, Pioneer Park of Lone Tree, Colonial Manor of the Columbus Community, Sunrise Terrace Nursing and Rehabilitation Center Parkview Home-Wayland.
* age 21-120

Exclusion criteria:

Only those who do not sign the consent form will be excluded

Exclusion Criteria:

* not a resident or primary care worker in one of the above listed retirement homes
* age less than 21 or greater than 110

Ages: 21 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2014-06; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Plaque index | 6 months
  Percentage reflecting the proportion of teeth surfaces covered by plaque, assessed by intra-oral exam.
Denture plaque index | 6 months
  Index reflecting the proportion of denture surfaces covered by plaque, assessed by denture exam.
Gingival bleeding index | 6 months
  Index reflecting the proportion of gingival areas Bleeding on probing, assessed by intra-oral exam.
Decayed, missing or filled surfaces (DMFS) index | 6 months
  Index reflecting the number of decayed, missing or filled teeth surfaces, assessed by intra-oral exam.
Total microbial count | 6 months
  Numbers of viable bacteria per swab will be determined following sector counting and analysis following standard spiral plating methodology
Isolation and enumeration of our target species: Porphyromonas gingivalis, Prevotella intermedia, Methicillin-Resistant Staphylococcus aureus (MRSA), Pseudomonas aeruginosa, Actinomyces spp., Fusobacterium nucleatum, and Candida albicans. | 6 months
  Plates will be counted following standard incubation times for each group of organisms and numbers of viable bacteria per swab will be determined following sector counting and analysis following standard spiral plating methodology.

SECONDARY OUTCOMES:
Assessment of residents cognitive status using Mini Cog test | 6 months
  Mini-Cog test is a 3-minute instrument to screen for cognitive impairment in older adults in the primary care setting.The instruments will be applied at baseline and end of the experiment protocol.
Assessment of cognitively sound participants quality of life using SF-36 questionnaire | 6 months
  The Short Form (36) Health Survey is a 36-item, patient-reported survey about quality of life. The instruments will be applied at baseline and end of the experiment protocol.
Assessment of cognitively sound participants oral health-related quality of life using OHIP 14 | 6 months
  Oral Health Impact Profile 14 questions questionnaire (OHIP-14) is a validated, commonly used, comprehensive questionnaire about oral-health related quality of life. The instruments will be applied at baseline and end of the experiment protocol.
Assessment of cognitively sound geriatric participants oral health-related quality of life using GOHAI | 6 months
  The Geriatric Oral Health Assessment Index (GOHAI) is a validated, widely used questionnaire developed to assess oral health perceptions among geriatric populations.The instruments will be applied at baseline and end of the experiment protocol.
Assessment of participants nutritional status using Mini Nutritional Assessment Short Form | 6 months
  The Mini Nutritional Assessment Short Form is a short questionnaire that also considers the BMI (weight in kg/height in m2) and provides an estimate of an individuals nutritional state. The instruments will be applied at baseline and end of the experiment protocol.
Assessment of number of events of x-ray documented pneumonia | 6 months
  X-ray documented pneumonia events are assessed through medical records at baseline and end of the experiment protocol.
Assessment of number of febrile days | 6 months
  Number of febrile days are assessed through medical records at baseline and end of the experiment protocol.
Assessment of dry mouth sensation | 6 months
  Participants are asked about feeling their mouth dry at baseline and by the end of the experimental protocol
Assessment of the presence of oral lesions | 6 months
  Presence of oral lesions was assessed by clinical exam at baseline and by the end of the experimental protocol

CONTACTS AND LOCATIONS:
Overall Officials: Brad Amendt, MS, Study Director — UIowa College of Dentistry
Locations (1):
- UIowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Undecided